CLINICAL TRIAL: NCT05713916
Title: A Pragmatic Clinical Trial Assessing the Effect of a Targeted Notification and Clinical Support Pathway on the Diagnostic Evaluation and Treatment of Individuals With Left Ventricular Hypertrophy
Brief Title: Effect of a Targeted Notification and Clinical Support Pathway on Individuals With Left Ventricular Hypertrophy
Acronym: NOTIFY-LVH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jason H. Wasfy, M.D.,M.Phil., Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022P002383
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hypertrophy, Left Ventricular; Hypertension; Cardiomyopathies
Keywords: Left ventricular hypertrophy; Pragmatic clinical trial
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Hypertension; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: Randomized pragmatic clinical trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Population Health Coordinator (Experimental): For subject randomized to the intervention arm, population health coordinators will notify the established longitudinal specialty clinician (cardiologist or nephrologist) or the primary care provider (PCP) that their patient has a recent echocardiogram demonstrating left ventricular hypertrophy (LVH). The outpatient clinician will be notified via the electronic health record (EHR) messaging system that the finding of LVH -- in the absence of significant valvular heart disease or a previously diagnosed cardiomyopathy -- may reflect undiagnosed or untreated hypertension.
  Interventions: Other: Intervention: Population Health Coordinator
- Observation: Usual Care (No Intervention): Those subjects randomized to the observation arm will receive usual care and their clinicians will not be notified about the finding of LVH on a prior echocardiogram until after study completion.

INTERVENTIONS:
Other: Intervention: Population Health Coordinator — After being notified of the finding of LVH in their patient, the population health coordinator will offer to schedule a dedicated visit for the provider and their patient to discuss this finding through a structured correspondence. Additionally, the population health coordinator will offer to coordinate 24-hour ambulatory blood pressure monitoring before or after the patient visit as part of the evaluation of LVH. Finally, for patients without established cardiovascular care and whose etiology of LVH remains undetermined, the population health coordinator will offer to coordinate a visit with a cardiologist to discuss the finding of LVH.
  Arms: Intervention: Population Health Coordinator

SUMMARY:
The electronic health record contains vast amounts of cardiovascular data, including potential clues that an individual may have unrecognized cardiac conditions. One important example is the finding of thickened heart muscle -- known as left ventricular hypertrophy (LVH) -- on echocardiograms (heart ultrasounds). If the underlying cause of LVH is untreated, individuals are at an increased risk of developing more severe pathology.

As the most common cause of LVH, hypertension and its downstream consequences account for more cardiovascular deaths than any other modifiable risk factor. Critically, many individuals have signs of cardiac damage from hypertension before it is diagnosed or treated. Despite this evidence, there are often gaps in healthcare delivery that contribute to substandard recognition and treatment. Thus, there is an urgent need to validate alternative cost-effective screening and intervention strategies.

Echocardiograms are ordered by many specialties and for numerous indications. Even when LVH is reported, the finding may be underappreciated and not prompt further evaluation. Whether data from prior echocardiograms can be harnessed to improve patient care through a centralized intervention is unknown.

Accordingly, the goal of this randomized pragmatic clinical trial is to study the impact of a centralized clinical support pathway on the diagnosis and treatment of hypertension and the recognition of LVH-associated diseases in individuals with evidence of thickened heart muscle on previously performed echocardiograms.

DETAILED DESCRIPTION:
The main questions our trial aims to answer are:

1. Can a centralized intervention designed to support and alert clinicians to the presence of LVH in their patients who are not being treated with blood pressure medications increase the diagnosis and treatment of hypertension?
2. Can a centralized clinical support intervention aimed at thoroughly screening for hypertension in individuals with LVH lead to an increase in the diagnosis of other causes of thickened heart muscle such as infiltrative and genetic cardiomyopathies?

For subjects randomized to the intervention arm, centralized population health coordinators will notify the established longitudinal specialty provider (cardiologist or nephrologist) or the primary care physician (PCP) that their patient has a recent echocardiogram demonstrating LVH. The outpatient clinician will be notified via the electronic health record messaging system that the finding of LVH -- in the absence of significant valvular heart disease or a previously diagnosed cardiomyopathy -- may reflect undiagnosed or untreated hypertension. Through a structured correspondence with the identified clinician, the population health coordinator will offer to schedule a dedicated visit for the provider and their patient to discuss the finding of LVH. Additionally, the population health coordinator will offer to coordinate 24-hour ambulatory blood pressure monitoring before or after the patient visit as part of the evaluation of LVH. Finally, for subjects without established cardiovascular care and whose etiology of LVH remains undetermined, the population health coordinator will offer to coordinate a visit with a cardiologist to discuss the finding of LVH.

Researchers will compare subjects randomized to the intervention arm against those randomized to the observation arm to determine if there are: (1) higher rates of initiation of blood pressure medications, (2) increased diagnoses of hypertension, and (3) increased diagnoses of alternate causes of thickened heart muscle in subjects randomized to the intervention arm of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-75 years
2. Transthoracic echocardiogram as of 1/1/2019
3. LVH on echocardiogram
4. Mass General Brigham PCP affiliation with at least 1 PCP practice visit within the last 24 months

Exclusion Criteria:

1. Current or previous outpatient blood pressure medication prescription
2. Moderate or severe aortic stenosis
3. Severe concentric LVH
4. Asymmetric LVH
5. History of prosthetic heart valve
6. Bicuspid aortic valve
7. Known cardiomyopathy (or had an outpatient visit diagnosis for a cardiomyopathy)
8. Autonomic dysfunction
9. History of heart or lung transplantation
10. Active cancer treatment plan
11. Active pregnancy
12. Dementia
13. Individuals whose primary address is in a nursing home or long-term care facility

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who are initiated on an antihypertensive medication | 12 months from the start of follow-up
  Collected from electronic health record data based on electronic prescribing data

SECONDARY OUTCOMES:
Number of participants who receive new diagnoses of hypertension | 12 months from the start of follow-up
  Collected from electronic health record data
Number of participants who are diagnosed with alternate causes of LVH (e.g., infiltrative cardiomyopathy, hypertrophic cardiomyopathy, etc.) that were not previously identified | 12 months from the start of follow-up
  Collected from electronic health record data

CONTACTS AND LOCATIONS:
Overall Officials: Jason H Wasfy, MD, Principal Investigator — Massachussets General Hospital; Adam N Berman, MD, Study Director — Brigham and Women's Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
After study completion, we will make every effort to make de-identified subject-level data available to other researchers upon reasonable request.
  Individual patient data that will be available upon reasonable request will include data that are presented in our study's main publication.
Supporting Information: Study Protocol, SAP
Time Frame: Individual patient data (de-identified) will made available upon reasonable request 6 months after publication of the trial's main findings.
Access Criteria: Researchers who request access to individual (de-identified) patient data may need to proceed with a formal Data Use Agreement through the Mass General Brigham Institutional Review Board.

REFERENCES:
- [Background] Cheng S, Claggett B, Correia AW, Shah AM, Gupta DK, Skali H, Ni H, Rosamond WD, Heiss G, Folsom AR, Coresh J, Solomon SD. Temporal trends in the population attributable risk for cardiovascular disease: the Atherosclerosis Risk in Communities Study. Circulation. 2014 Sep 2;130(10):820-8. doi: 10.1161/CIRCULATIONAHA.113.008506. Epub 2014 Aug 11. PMID 25210095
- [Background] Sakhuja S, Colvin CL, Akinyelure OP, Jaeger BC, Foti K, Oparil S, Hardy ST, Muntner P. Reasons for Uncontrolled Blood Pressure Among US Adults: Data From the US National Health and Nutrition Examination Survey. Hypertension. 2021 Nov;78(5):1567-1576. doi: 10.1161/HYPERTENSIONAHA.121.17590. Epub 2021 Oct 13. PMID 34644171
- [Background] Washington AE, Coye MJ, Boulware LE. Academic Health Systems' Third Curve: Population Health Improvement. JAMA. 2016 Feb 2;315(5):459-60. doi: 10.1001/jama.2015.18550. No abstract available. PMID 26836726
- [Background] Scirica BM, Cannon CP, Fisher NDL, Gaziano TA, Zelle D, Chaney K, Miller A, Nichols H, Matta L, Gordon WJ, Murphy S, Wagholikar KB, Plutzky J, MacRae CA. Digital Care Transformation: Interim Report From the First 5000 Patients Enrolled in a Remote Algorithm-Based Cardiovascular Risk Management Program to Improve Lipid and Hypertension Control. Circulation. 2021 Feb 2;143(5):507-509. doi: 10.1161/CIRCULATIONAHA.120.051913. Epub 2020 Nov 17. No abstract available. PMID 33201729
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2018 Oct 23;138(17):e484-e594. doi: 10.1161/CIR.0000000000000596. No abstract available. PMID 30354654
- [Background] Berman AN, Ginder C, Sporn ZA, Tanguturi V, Hidrue MK, Shirkey LB, Zhao Y, Blankstein R, Turchin A, Wasfy JH. Natural Language Processing for the Ascertainment and Phenotyping of Left Ventricular Hypertrophy and Hypertrophic Cardiomyopathy on Echocardiogram Reports. Am J Cardiol. 2023 Nov 1;206:247-253. doi: 10.1016/j.amjcard.2023.08.109. Epub 2023 Sep 13. PMID 37714095
- [Background] Berman AN, Ginder C, Wang XS, Borden L, Hidrue MK, Searl Como JM, Daly D, Sun YP, Curry WT, Del Carmen M, Morrow DA, Scirica B, Choudhry NK, Januzzi JL, Wasfy JH. A pragmatic clinical trial assessing the effect of a targeted notification and clinical support pathway on the diagnostic evaluation and treatment of individuals with left ventricular hypertrophy (NOTIFY-LVH). Am Heart J. 2023 Nov;265:40-49. doi: 10.1016/j.ahj.2023.06.014. Epub 2023 Jul 14. PMID 37454754
- [Derived] Berman AN, Hidrue MK, Ginder C, Shirkey L, Kwatra J, O'Kelly AC, Murphy SP, Searl Como JM, Daly D, Sun YP, Curry WT, Del Carmen MG, Blankstein R, Dodson JA, Morrow DA, Scirica BM, Choudhry NK, Januzzi JL Jr, Wasfy JH. Leveraging Preexisting Cardiovascular Data to Improve the Detection and Treatment of Hypertension: The NOTIFY-LVH Randomized Clinical Trial. JAMA Cardiol. 2025 Jul 1;10(7):686-695. doi: 10.1001/jamacardio.2025.0871. PMID 40162953